CLINICAL TRIAL: NCT03029377
Title: Noradrenergic and Stress-Related Etiologies of Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Gordon Bernard, Executive Vice President for Research, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 161423
Record Dates: First submitted 2017-01-09; First posted 2017-01-24 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Chronic Fatigue Syndrome
Keywords: CFS; Stress; Norepinephrine Transporter (NET); Norepinephrine (NE); Healthy Controls; Fatigue
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Fatigue Patients (Experimental): Patients between 18-60 years of age with fatigue symptoms who meet preliminary chronic fatigue phenotype criteria and complete preliminary screening surveys. Participants will undergo a Posture Study, Autonomic Function Tests, and a Stress Test. Participants' blood will be drawn to measure markers of sympathetic nervous system function.
  Interventions: Other: Posture Study, Autonomic Function Tests, and a Stress Test
- Healthy Controls (Active Comparator): Patients between 18-60 years of age with no known conditions or prescription medications who meet preliminary screening criteria. Participants will undergo a Posture Study, Autonomic Function Tests, and a Stress Test. Participants' blood will be drawn to measure markers of sympathetic nervous system function.
  Interventions: Other: Posture Study, Autonomic Function Tests, and a Stress Test

INTERVENTIONS:
Other: Posture Study, Autonomic Function Tests, and a Stress Test — Participants will undergo a Posture Study, Autonomic Function Tests, and a Stress Test. Participants' blood will be drawn to measure markers of sympathetic nervous system function at baseline, in three postural positions, after autonomic tests, and after a stress test.

SUMMARY:
The objective of this study is to measure sympathetic nervous system function and stress responses in patients with clinically documented and self-reported chronic fatigue that is worsened by stress, compared to healthy controls. Baseline norepinephrine (NE) levels and stress-induced NE levels in patients who fulfill criteria for Chronic Fatigue Syndrome (CFS) and who self-identify with stress induced worsening fatigue, will be compared to data from normal individuals pre and post-stress.

DETAILED DESCRIPTION:
Symptoms of Chronic Fatigue Syndrome (CFS) are critically important to study as patients report that these symptoms are often profoundly debilitating and an impediment to effective daily functioning as well as effective vocational and social functioning, while also contributing to a significantly increased risk of psychiatric illness and diminished quality of life. Previous Phenome-Wide Association (PheWAS) studies revealed a link between a norepinephrine transporter (NET) genetic variant and CFS. Based on the potential function of the variant and published literature, elevated norepinephrine (NE) levels may underlie at least some cluster of fatigue symptoms. Some patients may experience chronic fatigue that is due to an excess of circulating NE, and fatigue symptoms are reported by our patient population to be commonly exacerbated by stress. This study will test the hypothesis that in a subset of people with severely debilitating fatigue of long duration (>6 months) that is worsened by stress identified through the Vanderbilt electronic health record phenotyping study, have chronic over-release of the hormone NE into the bloodstream/periphery over time that results in an overload of NE. This overload of NE causes a compensatory but deleterious effect on the brain and nervous system, including sympathetic effects and dysregulated physiologic response to stress. Thus, while numerous currently approved therapies that target NET inhibit the transporter, a drug with the opposite mechanism of action, a NET activator that would decrease circulating NE, may have efficacy in treating underlying pathophysiology of chronic fatigue.

Baseline NE levels and stress-induced NE levels in patients who fulfill criteria for CFS and who self-identify with stress induced worsening fatigue, will be compared to data from normal individuals pre and post-stress. After all inclusion criteria has been confirmed, an IV will be placed for blood collection, a continuous electrocardiographic trace and blood pressure cuff will be placed on the subject's arm and finger. Subjects will undergo a posture study, autonomic reflex testing, and Stroop stress testing each followed by blood specimen collection. An optional blood draw for DNA analysis will occur after patients have been provided lunch. Questionnaires will be completed after study procedures and patients have been provided lunch. Study blood collection will total up to 28 milliliters (mL): 5 mL for cytokines, 20 mL for catecholamines, and optional 3 mL for DNA.

ELIGIBILITY:
Chronic Fatigue Participants:

Inclusion Criteria:

* Confirmed chronic fatigue with severity >50 on a scale of 1 to 100 that is not improving over time
* Meet The Centers for Disease Control and Prevention (CDC) diagnostic criteria of CFS (self-reported persistent or relapsing fatigue lasting 6 or more consecutive months)

Exclusion Criteria:

* Male and female subjects <18 or >60 years
* Obesity, defined as a BMI of 30 or more
* Presence of other medical or psychiatric conditions known to cause fatigue (alcohol/drug abuse, anorexia nervosa, bipolar disorder, bulimia nervosa, dementia, major depression, psychotic/delusional disorders, schizophrenia)
* Presence of sleep disorder/disruption known to cause fatigue (sleep apnea, narcolepsy)
* Cardiovascular, pulmonary, hepatic, or hematological disease by history or prior testing defined as significant by investigator (including but not limited to chronic hepatitis, chronic kidney disease, cirrhosis, emphysema, heart failure, HIV, lupus, multiple sclerosis, myasthenia gravis, rheumatoid arthritis)
* History of hypertension defined as supine resting BP>145/95 mmHg off medications or needing antihypertensive medication
* Patients taking medications that can affect autonomic function or plasma catecholamines (vasoactive drugs), stimulants, and/or are sedatives
* Other factors which in the opinion of the investigator could potentially impact the study outcomes (e.g., underlying disease, medications, history)* or prevent the participant from completing the protocol (poor compliance or unpredictable schedule)
* Inability to stand unassisted for 10 minutes
* Patients who are bedridden or chair-ridden
* Patients who are colorblind
* Inability or refusal to give informed consent for any reason including a diagnosis of dementia or cognitive impairment
* Patients who are pregnant or breastfeeding

Healthy Control Participants:

* Participant with no significant reported conditions or medications.

Exclusion Criteria:

* Male and female subjects <18 or >60 years
* Obesity, defined as a BMI of 30 or more
* Presence of any serious or chronic disease, or prescription medication as deemed by investigator including hypertension as defined by supine resting BP >145/95 mmHg off medications or needing antihypertensive medication
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule
* Inability to stand unassisted for 10 minutes
* Patients who are bedridden or chair-ridden
* Patients who are colorblind
* Inability or refusal to give informed consent for any reason including a diagnosis of dementia or cognitive impairment
* Patients who are pregnant or breastfeeding
* Stress Overload Score above 66

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
dihydroxyphenylglycol (DHPG)/norepinephrine (NE) Ratio (post stress) | Change from Baseline to post stress test (approximately 100 minutes post-baseline blood collection)
  Change in DHPG/NE Ratio from Baseline to post stress compared across arms

SECONDARY OUTCOMES:
DHPG/NE Ratio (post Autonomic Function test) | Change from Baseline to post Autonomic Function test (approximately 30 minutes post-baseline blood collection)
  Change in DHPG/NE Ratio from Baseline to post Autonomic Function test compared across arms
DHPG/NE Ratio (post Standing position) | Change from Baseline to post Standing position (approximately 40 minutes post-baseline blood collection)
  Change in DHPG/NE Ratio from Baseline to post Standing position compared across arms
DHPG/NE Ratio (post Sitting position) | Change from Baseline to post Sitting position (approximately 70 minutes post-baseline blood collection)
  Change in DHPG/NE Ratio from Baseline to post Sitting position compared across arms
Absolute DHPG and NE Levels (post stress) | Change from Baseline to post stress test (approximately 100 minutes post-baseline blood collection)
  Change in absolute DHPG and NE Levels from Baseline to post stress compared across arms
Absolute DHPG and NE Levels (post Autonomic Function test) | Change from Baseline to post Autonomic Function test (approximately 30 minutes post-baseline blood collection)
  Change in DHPG and NE levels from Baseline to post Autonomic Function test compared
Absolute DHPG and NE Levels (post Standing position) | Change from Baseline to post Standing position (approximately 40 minutes post-baseline blood collection)
  Change in absolute DHPG and NE Levels from Baseline to post Standing position compared across arms
Absolute DHPG and NE Levels (post Sitting position) | Change from Baseline to post Sitting position (approximately 70 minutes post-baseline blood collection)
  Change in DHPG and NE levels from Baseline to post Sitting position compared across arms
Fatigue as assessed by Multidimensional Assessment of Fatigue Scale (MAF) | End of Study Visit (approximately 140 minutes post-baseline blood collection)
  Mean values +/- standard deviation (SD) compared across arms
Mood as assessed by Hospital Anxiety and Depression Scale (HADS) | End of Study Visit (approximately 140 minutes post-baseline blood collection)
  Mean values +/- SD compared across arms
Quality of Life as assessed by 36-Item Short Form Survey Instrument (SF-36) | End of Study Visit (approximately 140 minutes post-baseline blood collection)
  Mean values +/- SD compared across arms
Stress as assessed by Stress Overload Scale | Beginning of Study Visit (Approximately 15 minutes pre-baseline blood collection)
  Mean values +/- SD compared across arms
Cytokines | At baseline (approximately 30 minutes after supine position start)
  Compared across arms

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bernard, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okamoto LE, Raj SR, Peltier A, Gamboa A, Shibao C, Diedrich A, Black BK, Robertson D, Biaggioni I. Neurohumoral and haemodynamic profile in postural tachycardia and chronic fatigue syndromes. Clin Sci (Lond). 2012 Feb;122(4):183-92. doi: 10.1042/CS20110200. PMID 21906029
- [Background] Shirey-Rice JK, Klar R, Fentress HM, Redmon SN, Sabb TR, Krueger JJ, Wallace NM, Appalsamy M, Finney C, Lonce S, Diedrich A, Hahn MK. Norepinephrine transporter variant A457P knock-in mice display key features of human postural orthostatic tachycardia syndrome. Dis Model Mech. 2013 Jul;6(4):1001-11. doi: 10.1242/dmm.012203. Epub 2013 Apr 4. PMID 23580201
- [Background] Danciu I, Cowan JD, Basford M, Wang X, Saip A, Osgood S, Shirey-Rice J, Kirby J, Harris PA. Secondary use of clinical data: the Vanderbilt approach. J Biomed Inform. 2014 Dec;52:28-35. doi: 10.1016/j.jbi.2014.02.003. Epub 2014 Feb 14. PMID 24534443
- See also: CDC - Chronic Fatigue Syndrome (CFS) — http://www.cdc.gov/cfs/